CLINICAL TRIAL: NCT05197335
Title: Observational, Prospective and Multicentre Clinical Study for the Evaluation of Clinical Parameters of Elderly Patients With Fractures of the Proximal Femur Treated by the Intramedullary Nail Chimaera (Orthofix Srl) Italian on Documents: Indagine Clinica Osservazionale, Prospettica e Multicentrica Per la Valutazione di Parametri Clinici di Pazienti Anziani Con Frattura Del Femore Prossimale Trattata Mediante il Chiodo Intramidollare Chimaera (Orthofix Srl)
Brief Title: Observational Clinical Study on Elderly Patients With Fracture of the Proximal Femur Treated With the Chimaera Nail
Acronym: Chimaera
Status: Completed | Type: Observational
Sponsor: Orthofix s.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: OCI_1901
Record Dates: First submitted 2021-12-23; First posted 2022-01-19 (Actual); Results first posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Hip Fractures; Subtrochanteric Fractures; Intertrochanteric Fractures; Pertrochanteric Fracture
Keywords: Femur; Fracture; Femoral; Nail; Nailing; Trochanteric; Sliding; Screw; Intramedullary; Elderly Patients
MeSH Terms: conditions — Hip Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Age of 65 at the time of signing the informed consent.
  Interventions: Device: Chimaera short nail (length = 180 mm) in combination with one or two telescopic cephalic screws

INTERVENTIONS:
Device: Chimaera short nail (length = 180 mm) in combination with one or two telescopic cephalic screws — The enrolled patients will proceed by undergoing the surgery necessary for the application of the medical device under observation (Chimaera), which coincides with the start of the treatment period.

SUMMARY:
This is an observational, prospective and multicenter clinical investigation that is part of the active materiovigilance plan that Orthofix Srl, in agreement with its Notified Body. The sponsor has planned to actively collect clinical data relating to the use of Chimaera Intramedullary Nail in a representative number of users and elderly patients with fractures of the proximal femur. The data obtained from this clinical investigation will be used to complete the pre-market clinical evaluation carried out on the Chimaera with post-market clinical data from the use of the device in normal clinical practice.

DETAILED DESCRIPTION:
Orthofix Srl has developed and placed on the European market the Chimaera Intramedullary Nail after having evaluated the clinical performance and safety of the medical device based on biomechanical tests and clinical data obtained from scientific publications on equivalent products. The outcome of this pre-market assessment established that Chimaera possesses the requirements for CE marking, in particular, it possesses an acceptable risk/benefit ratio if used according to the manufacturer's directions for use.

The enrolled patients, as would happen even if they did not decide to participate in this study, will proceed by undergoing the surgery necessary for the application of the medical device under observation (Chimaera), which coincides with the start of the treatment period.

After the surgery and the hospital discharge, the patient will undergo subsequent follow-up visits. The follow-up visits carried out respectively at 1 month and 3 months after the date of surgery, conclude the treatment period which, barring complications, is expected within 8 - 12 weeks from the date of surgery with the consolidation of the fracture of the proximal femur treated. Healing will be verified by the Investigator based on an X-ray check through which he/she will make a qualitative assessment of the bone density at the fracture site and the positioning of the bone stumps. Starting from the 3-month visit and up to 1-year visit, the Investigator will compile the Bowers & Parker functional score (a measure of effectiveness) for the evaluation of the patient's functional recovery. The score obtained at the follow-up visits will be compared to the score compiled during the discharge visit representative of the pre-fracture patient's status.

For patients that undergo this treatment, the removal of the device is not planned except for serious adverse events that require a second surgery to complete the treatment of the fracture (safety measure). Once the treatment period has ended, the control period begins during which 2 visits will be made, respectively 6 months and 1 year after the date of the surgery. During these visits, clinical data will be collected to follow the evolution of the fracture consolidation and the functional recovery of the patient and the occurrence of any adverse events in the medium term.

ELIGIBILITY:
Inclusion Criteria:

* directly or indirectly (through a respondent) will have expressed their will to participate in the study by signing and dating the informed consent;
* will have reached the age of 65 at the time of signing the informed consent;
* he/she will have been diagnosed with a fracture in the pertrochanteric, intertrochanteric or subtrochanteric region of the femur, stable or unstable, not previously treated;
* based on the investigator's judgment, he will have a regular indication for surgical treatment with an intramedullary nail;
* the fracture will be treated with the Chimaera short nail (length = 180 mm) and one or two telescopic lag screws, according to the manufacturer's instructions for use.

Exclusion Criteria:

* will undergo surgery to treat the results of a previously treated fracture;
* he/she will have been diagnosed with a pathological fracture of oncological origin (primary tumor or skeletal metastasis);
* he/she will have been diagnosed with a fracture in the diaphyseal and/or distal region of the femur;
* he/she will have been diagnosed with an open fracture (type II and III according to the classification of Gustilo and Anderson) of the proximal femur;
* he/she will have been diagnosed with multiple fractures (including bilateral proximal femur fractures);
* in the pre-or intra-operative phase it will be decided to treat the fracture with the long version of the Chimaera nail and/or with non-telescopic cephalic screws (fixed length);
* will have a medical condition that constitutes a contraindication to treatment with Chimaera according to the manufacturer's instructions for use;
* will have a suspected or certified hypersensitivity/allergy to some component of the device that comes into contact with the patient;
* will present some clinical condition that, in the Investigator's opinion, could interfere with the procedures of the Clinical Investigation or that could jeopardize the safety of the patient;
* at the same time he will be treated with an unauthorized device that cannot be removed without endangering the safety of the patient;
* will be participating in other clinical trials or had participated in other clinical trials in the 3 months before signing the informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: An adult patient with a previously untreated proximal femur fracture who, based on the free judgment of the Investigator, will have a regular indication for surgical treatment with Chimaera will be considered eligible for participation in the clinical investigation. Eligible patients who meet the inclusion criteria and no exclusion criteria will be considered eligible for participation in this Clinical Investigation.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - Ospedale Regionale EE 'Miulli', Acquaviva delle Fonti, BA
  - A.O. Sant'Anna e San Sebastiano Caserta, Caserta, CE
  - A.O.U. Policlinico - Vittorio Emanuele, Catania, CT
  - Ospedale S. Giuseppe, Empoli, FI
  - Az. Ospedaliero - Universitaria Careggi, Florence, FI
  - ASST di Mantova, Osp. Carlo Poma, Mantova, MN
  - Nuovo Ospedale di Prato S. Stefano, Prato, PO
  - Ospedale di Vicenza, Vicenza, VI

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Close JD, Swartz K, Deu R. Hip fracture in older patients: tips and tools to speed recovery. J Fam Pract. 2013 Sep;62(9):484-92. PMID 24080557
- [Background] Sheehan SE, Shyu JY, Weaver MJ, Sodickson AD, Khurana B. Proximal Femoral Fractures: What the Orthopedic Surgeon Wants to Know. Radiographics. 2015 Sep-Oct;35(5):1563-84. doi: 10.1148/rg.2015140301. Epub 2015 Jul 17. PMID 26186669
- [Background] Innocenti M, Civinini R, Carulli C, Matassi F. Proximal femural fractures: epidemiology. Clin Cases Miner Bone Metab. 2009 May;6(2):117-9. PMID 22461159
- [Background] Orive M, Aguirre U, Garcia-Gutierrez S, Las Hayas C, Bilbao A, Gonzalez N, Zabala J, Navarro G, Quintana JM. Changes in health-related quality of life and activities of daily living after hip fracture because of a fall in elderly patients: a prospective cohort study. Int J Clin Pract. 2015 Apr;69(4):491-500. doi: 10.1111/ijcp.12527. Epub 2015 Feb 27. PMID 25721490
- [Background] Sciard D, Cattano D, Hussain M, Rosenstein A. Perioperative management of proximal hip fractures in the elderly: the surgeon and the anesthesiologist. Minerva Anestesiol. 2011 Jul;77(7):715-22. Epub 2011 Feb 1. PMID 21283071
- [Background] Prestmo A, Hagen G, Sletvold O, Helbostad JL, Thingstad P, Taraldsen K, Lydersen S, Halsteinli V, Saltnes T, Lamb SE, Johnsen LG, Saltvedt I. Comprehensive geriatric care for patients with hip fractures: a prospective, randomised, controlled trial. Lancet. 2015 Apr 25;385(9978):1623-33. doi: 10.1016/S0140-6736(14)62409-0. Epub 2015 Feb 5. PMID 25662415
- [Background] Bowers TM, Parker MJ. Assessment of outcome after hip fracture: development of a universal assessment system for hip fractures. SICOT J. 2016;2:27. doi: 10.1051/sicotj/2016018. Epub 2016 Jun 3. PMID 27259572
- See also: ICJME. Recommendations for the Conduct, Reporting, Editing, and Publication of Scholarly work in Medical Journals. — http://www.icmje.org/recommendations/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Group
Started | 206
Completed | 131
Not Completed | 75

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 206
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 84.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 206
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 206

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Needing a Second Surgery
Description: Safety measurement outcome: the percentage of patients who, due to serious adverse events related to Chimaera, will have to undergo a second surgery to continue with the treatment of the proximal femur fracture.
Time Frame: 6 months
Population: Adult patients with a previously untreated proximal femur fracture who, in the Investigator's sole judgment, has a standard indication for surgical treatment with Chimaera will be considered eligible for participation in the clinical investigation. Eligible patients who meet the following inclusion criteria and none of the exclusion criteria will be considered suitable for participation in this Clinical Investigation.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 206
Participants | 0

2. Secondary Outcome: Functional Score of Bowers & Parker
Description: Efficacy measurement outcome: the functional score of Bowers & Parker for the evaluation of the functional recovery of the patient. This score is made of three continuous scales defined for pain, mobility and functional independence. The Pain score is assessed from 0 (Unable to answer) to 8 (Constant and severe pain in the hip requiring regular strong analgesia such as opiates). The Mobility score is assessed from 1 (Never uses any walking aid and no restriction in walking distance) to 10 (Bedbound most or all of the day). The Functional score is assessed from 1 (Completely independent. Requires no assistance in basic or advanced activities of daily living (ADL) including shopping) to 8 (Patient temporarily resident in hospital requiring both nursing and medial care).
Time Frame: 12 months
Population: Adult patients with a previously untreated proximal femur fracture who, in the Investigator's sole judgment, has a standard indication for surgical treatment with Chimaera will be considered eligible for participation in the clinical investigation. We report the Bowers & Parker functional score results at one year after surgery (Visit 6), based on data from 129 patients who completed the assessment at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 129
score on a scale
  Mobility | 4.11 (2.49)
  Independence | 3.14 (1.75)
  Pain | 1.73 (1.36)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the postoperative follow-up period of up to 6 months. The safety of the Chimaera device was assessed based on the percentage of patients who required a second surgical procedure due to serious adverse events related to the device.
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 28/206
Serious Adverse Events (participants affected / at risk) | 79/206
Other Adverse Events (participants affected / at risk) | 23/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=206)
Postoperative anemia (Injury, poisoning and procedural complications) | 14 (14)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Fracture and Fall (Injury, poisoning and procedural complications) | 1 (1)
Death (General disorders) | 22 (22)
Disease complication and Peripheral oedema peripheral (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 8 (8)
Endocarditis (Infections and infestations) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 4 (4)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Delirium (Nervous system disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Marasmus (Metabolism and nutrition disorders) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Red blood cell transfusion (Surgical and medical procedures) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=206)
Urinary Infection (Infections and infestations) | 6 (6)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 5 (5)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2)
Oedema peripheral (General disorders) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT05197335/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT05197335/ICF_001.pdf